CLINICAL TRIAL: NCT04963504
Title: Pulmonary Diffusing Capacity Changes to Posture and Acute Exercise in Healthy Volunteers: a Randomised Test-retest Relaibility Study
Brief Title: Pulmonary Diffusing Capacity During Postural Postural Changes and Acute Exercise
Acronym: DiffLung
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Ronan Berg, Associate Professor, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KF_458_21
Record Dates: First submitted 2021-07-05; First posted 2021-07-15 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Clinical Assessments of Pulmonary Diffusing Capacity

STUDY DESIGN:
Intervention Model Description: Randomised study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rest-to-exercise (Experimental)
  Interventions: Diagnostic Test: Rest-to-exercise
- Sitting-to-supine (Experimental)
  Interventions: Diagnostic Test: Sitting-to-supine

INTERVENTIONS:
Diagnostic Test: Rest-to-exercise — Pulmonary diffusing capacity is assessed at rest and during exercise (70% of VO2max on a bicycle ergometer)
  Arms: Rest-to-exercise
Diagnostic Test: Sitting-to-supine — Pulmonary diffusing capacity is assessed in the sitting and supine position
  Arms: Sitting-to-supine

SUMMARY:
The combined measurement of the pulmonary diffusing capacity to carbon monoxide (CO) and nitric oxide (NO) (DLCO/NO) has recently been standardised and validated for clinical use. It involves a very short breath-hold time (≤5 seconds), and it may be repeated up to 12 times without affecting measurements, and it is thus ideal for assessing acute changes in pulmonary diffusing capacity and its components during various physiological manoeuvres. The aim of the present study is to compare the test-retest reliability of pulmonary diffusing capacity measurements during postural changes (sitting vs. supine) vs. rest-to-exercise. DLCO/NO will either be measured in the sitting position during rest vs. exercise or in the sitting and supine posture, and this will be repeated within 1-7 days in 20 healthy individuals that will be randomised to one of the two interventions. Statistically,the test-retest relaibility of sitting-to-supine vs. rest-to-exercise changes in DLCO/NO will be compared by parametric methods.

ELIGIBILITY:
Inclusion Criteria:

• Regular exercise (1-3 timer per week)

Exclusion Criteria:

* Any known medical condition that requires regular medication or any known lung condition
* Smoking
* Symptoms of disease within 2 weeks prior to the study
* Abnormal lung function test
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Between intervention DLNO/DLCO-ratio repeatability coefficient | 1 week
  Test-retest reliability coefficient of rest-to-exercise and supine-to-prone DLNO/DLCO-ratio
Between intervention DLCO repeatability coefficient | 1 week
  Test-retest repeatability coefficient of rest-to-exercise and supine-to-prone DLCO
Between intervention DLNO repeatability coefficient | 1 week
  Test-retest repeatability coefficient of rest-to-exercise and supine-to-prone DLNO

SECONDARY OUTCOMES:
Between intervention DM repeatability coefficient | 1 week
  Test-retest repeatability coefficient of rest-to-exercise and supine-to-prone DM
Between intervention Vc repeatability coefficient | 1 week
  Test-retest repeatability coefficient of rest-to-exercise and supine-to-prone Vc

OTHER OUTCOMES:
Between day DLNO/DLCO-ratio repeatability coefficient | 1 week
  Between-day repeatability coefficient of DLNO/DLCO at rest in both groups combined
Between day DLCO repeatability coefficient | 1 week
  Between-day repeatability coefficient of DLCO at rest in both groups combined
Between day DLNO repeatability coefficient | 1 week
  Between-day repeatability coefficient of DLNO at rest in both groups combined
Between day DM repeatability coefficient | 1 week
  Between-day repeatability coefficient of DM at rest in both groups combined
Between day Vc repeatability coefficient | 1 week
  Between-day repeatability coefficient of Vc at rest in both groups combined
DLNO/DLCO-ratio MDC | 1 week
  Between-day MDC of DLNO/DLCO from rest-to-exercise and supine-to-prone
DLCO MDC | 1 week
  Between-day MDC of DLCO from rest-to-exercise and supine-to-prone
DLNO MDC | 1 week
  Between-day MDC of DLNO from rest-to-exercise and supine-to-prone
DM MDC | 1 week
  Between-day MDC of DM from rest-to-exercise and supine-to-prone
Vc MDC | 1 week
  Between-day Vc of DM from rest-to-exercise and supine-to-prone
DLNO/DLCO-ratio ICC | 1 week
  Between-day ICC of DLNO/DLCO from rest-to-exercise and supine-to-prone
DLCO ICC | 1 week
  Between-day ICC of DLCO from rest-to-exercise and supine-to-prone
DLNO ICC | 1 week
  Between-day ICC of DLNO from rest-to-exercise and supine-to-prone
DM ICC | 1 week
  Between-day ICC of DM from rest-to-exercise and supine-to-prone
Vc ICC | 1 week
  Between-day ICC of Vc from rest-to-exercise and supine-to-prone
DLNO/DLCO-ratio SEM | 1 week
  Between-day SEM of DLNO/DLCO from rest-to-exercise and supine-to-prone
DLCO SEM | 1 week
  Between-day SEM of DLCO from rest-to-exercise and supine-to-prone
DLNO SEM | 1 week
  Between-day SEM of DLNO from rest-to-exercise and supine-to-prone
DM SEM | 1 week
  Between-day SEM of DM from rest-to-exercise and supine-to-prone
Vc SEM | 1 week
  Between-day SEM of Vc from rest-to-exercise and supine-to-prone
DLNO/DLCO-ratio CV | 1 week
  Between-day CV of DLNO/DLCO from rest-to-exercise and supine-to-prone
DLCO CV | 1 week
  Between-day CV of DLCO from rest-to-exercise and supine-to-prone
DLNO CV | 1 week
  Between-day CV of DLNO from rest-to-exercise and supine-to-prone
DM CV | 1 week
  Between-day CV of DM from rest-to-exercise and supine-to-prone
Vc CV | 1 week
  Between-day CV of Vc from rest-to-exercise and supine-to-prone

CONTACTS AND LOCATIONS:
Overall Officials: Ronan Berg, MD, Principal Investigator — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be shared upon reasonable request.